CLINICAL TRIAL: NCT05837052
Title: A Phase II Trial to Evaluate the Efficiency and Safety of Serplulimab Plus Chemotherapy as Conversion Treatment for Patients With Stage IIIB-IVA Oligometastatic Non-small Cell Lung Cancer
Brief Title: A Phase II Trial to Evaluate the Efficiency and Safety of Serplulimab Plus Chemotherapy as Conversion Therapy in NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Weijia Fang, MD, Professor, Zhejiang University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTHLX10
Record Dates: First submitted 2023-04-17; First posted 2023-05-01 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Unresectable Lung Non-Small Cell Carcinoma
Keywords: Unresectable NSCLC; Serplulimab; Conversion treatment
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serplulimab plus chemotherapy (Experimental): Patients with unresectable NSCLC will receive 3-4 cycles of serplulimab plus chemotherapy as the conversion treatment (serplulimab 300mg d1 q3w; carboplatin (AUC 5) on day 1, and pemetrexed (500 mg/m2 for adenocar- cinoma) or nab-paclitaxel (260 mg/m2 for squamous carcinoma) d1 q3w), and then curative pneumonectomy will be provided for patients who are suitable for primary tumor resection. Locoregional ablative treatments will be performed for metastatic lesions. Maintenance treatment with PD-1 antibody q3w will continue up to 12 months or disease progression after surgery.
  Interventions: Procedure: serplulimab plus chemotherapy as conversion treatment

INTERVENTIONS:
Procedure: serplulimab plus chemotherapy as conversion treatment — Patients with unresectable NSCLC will receive serplulimab plus chemotherapy as conversion treatment, and then curative pneumonectomy will be provided for patients who are suitable for primary tumor resection. Locoregional ablative treatments will be performed for metastatic lesions.

SUMMARY:
This is a phase II, single-arm study to evaluate the efficacy and safety of Serplulimab plus chemotherapy as conversion treatment in patients with stage IIIB-IVA oligometastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
This single-arm, open-label, prospective phase II clinical trial was designed to evaluate the efficacy and safety of Serplulimab plus chemotherapy as conversion treatment in patients with stage IIIB-IVA oligometastatic non-small cell lung cancer.

The primary endpoints were the rate of NSCLC converting to resectable tumors and the 1-year progression-free survival (PFS) rate.The secondary endpoints included the rates of R0 resection, major pathological response (MPR) and pathological complete response (pCR), overall survival (OS) and PFS. Multi-omics analysis will be performed to identify potential biomarkers for treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should voluntarily join this study and sign the informed consent form
2. NSCLC patients diagnosed by cytology or histology and not previously receiving anti-tumor treatments (including systemic treatments, local treatments .etc)
3. Patients with IIIB - IVA oligometastatic NSCLC : (a) IIIB - IIIC stage (T1-4N2-3): patients are not suitable or refuse to receive upfront surgical resection or radiotherapy; (b) oligometastatic stage IV (T1-3N0-2): radical resection/radiotherapy is feasible for metastatic lesions (the number of metastases being up to 3, and the maximum diameter of metastases being up to 2cm)
4. After evaluation by MDT, upfront surgical resection is not the preferred treatment, but after induction systemic treatments, radical resection of the primary tumor is feasible, and radical resection/radiotherapy is feasible for extrathoracic metastases (if any)
5. Age from 18 to 75 years old, both male and female
6. ECOG score 0-1
7. According to the RECIST v1.1 , patients should have at least one measurable lesion
8. For suspicious mediastinal lymph nodes (including pathological enlargement or PET-CT indicating malignancy, etc.), further sampling is required for pathological diagnosis by EUBS, thoracoscopy, or mediastinoscopy
9. According clinical evaluation, the lung function of patients (such as FVC, FEV1, TLC, FRC, DLco, etc.) should be sufficient for pneumonectomy
10. The function of important organs should meet the following requirements: absolute count of neutrophils ≥ 1.5 × 109/L； Platelets ≥ 100 × 109/L； Hemoglobin ≥ 90g/L; Serum albumin ≥ 35g/L; Thyroid hormone (TSH) ≤ 1 × ULN； Serum bilirubin ≤ 1.5 × ULN； ALT and AST ≤ 3 × ULN； International standardized ratio (INR) ≤ 1.5 or prothrombin time (PT) ≤ 1.5 × ULN； Serum creatinine ≤ 1.5 × ULN
11. Female patients at childbearing age are required to use contraceptive measures; for male patients whose partners are women at childbearing age, effective methods of contraception should be used during the trial period

Exclusion Criteria:

Patients who meet any of the following conditions will not be enrolled in this study:

1. NSCLC patients have sensitive EGFR mutation, EML4-ALK fusion or other forms of ALK gene changes
2. Patients have previously received immune checkpoint inhibitors such as PD-1/ PD-L1/CTLA4 antibody
3. Patients with other primary malignancies within the past 3 years (excluding cured skin basal cell carcinoma and cervical carcinoma in situ)
4. Patients with active hepatitis B/C
5. Patients with any active autoimmune diseases or a history of autoimmune diseases
6. Patients who are using immunosuppressive agents or require systemic hormone therapy
7. Patients with hypertension but without good control even through antihypertensive medication treatment ; patients with clinical symptoms or diseases related to unsatisfying cardiac function
8. Patients with abnormal coagulation function (INR>2.0, PT>16s)
9. Arterial/venous thrombotic events occurred before screening within 6 months
10. Patients with active infection
11. Patients with congenital or acquired immune dysfunction (such as HIV infection)
12. According to the judgment of the researchers, patients have other factors that may affect the results of the research or cause the research to be terminated

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
the rate of NSCLC converting to resectable tumors | up to 16 weeks
  the proportion of unresectable NSCLC patients who are converted to being suitable for radical pneumonectomy after 3-4 cycles serplulimab plus chemotherapy
the 1-year progression-free survival (PFS) rate | up to one year
  the proportion of patients who are progression-free after pneumonectomy

SECONDARY OUTCOMES:
the rate of R0 resection | immediately after the surgery
  the proportion of R0 resection in patients who receive pneumonectomy
Progression-free survival (PFS) | up to five years
  The duration from the date of initial treatment to the date of disease progression or death due to any cause
Overall survival (OS) | up to five years
  The duration from the date of initial treatment to the date of death due to any cause
the rate of major pathological response (MPR) | up to 16 weeks
  the proportion of patients who achieve MRP among those receiving pneumonectomy
the rate of pathological complete response (pCR) | up to 16 weeks
  the proportion of patients who achieve pCR among those receiving pneumonectomy

CONTACTS AND LOCATIONS:
Overall Officials: Weijia Fang, MD, Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (1):
- Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No